CLINICAL TRIAL: NCT00702026
Title: The Effect of a Multispecies Probiotic on Hypersensitivity in IBS Patients
Brief Title: The Effect of a Multispecies Probiotic on Hypersensitivity in Irritable Bowel Syndrome (IBS) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Winclove Bio Industries BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEC 08-1-031
Record Dates: First submitted 2008-06-11; First posted 2008-06-19 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Irritable Bowel Syndrome; Hypersensitivity
Keywords: Irritable Bowel Syndrome; Hypersensitivity; Probiotics; Multispecies
MeSH Terms: conditions — Irritable Bowel Syndrome; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: multispecies probiotic (Ecologic 801)
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: multispecies probiotic (Ecologic 801) — once daily, 5 gram [10e9 cfu/gram]
  Other Names: Ecologic 801
  Arms: 1
Dietary Supplement: Placebo — once daily, 5 gram [10e9 cfu/gram]
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether a specifically designed multispecies probiotic decreases visceral hypersensitivity in IBS-patient (defined by an increased pain tolerance threshold). Moreover, the effect on general symptom scores and inflammatory and microbiological parameters will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of IBS according to the Rome III criteria
* Increased visceral perception according to barostat measurements, defined as a pain tolerance threshold at smaller than or equal to 23 mmHg
* Age between 18 and 65 years
* BMI between 18.5 and 30 kg/m2

Exclusion Criteria:

* Known gastro-intestinal diseases
* Major abdominal surgery
* Previous radiotherapy, chemotherapy
* Clinical significant systemic diseases
* Critically ill patients or patients suffering from severe acute pancreatitis
* Patients with organs failure
* Patients receiving enteral feeding
* Excessive alcohol intake (greater than 15 consumptions per week)
* (planned) pregnancy or lactation
* Use of pre-, probiotics in the month before and during the study
* Use of antibiotics in the two months before and during the study
* Use of anti-diarrhoea medication, anti-laxatives or anti-acid medication in the two weeks before and during the study
* Use of anti depressives (especially SSRI's) in the month before and during the study
* Use of other medication if less then one month on stable dosage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain tolerance threshold | t=0 and t=6 weeks
VAS score for pain at pressure step 29 mmHg | t=0 and t=6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: A AM Masclee, Prof. Dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands

REFERENCES:
- [Derived] Ludidi S, Mujagic Z, Jonkers D, Keszthelyi D, Hesselink M, Kruimel J, Conchillo J, Masclee A. Markers for visceral hypersensitivity in patients with irritable bowel syndrome. Neurogastroenterol Motil. 2014 Aug;26(8):1104-11. doi: 10.1111/nmo.12365. Epub 2014 Jun 11. PMID 24920528
- [Derived] Ludidi S, Jonkers DM, Koning CJ, Kruimel JW, Mulder L, van der Vaart IB, Conchillo JM, Masclee AA. Randomized clinical trial on the effect of a multispecies probiotic on visceroperception in hypersensitive IBS patients. Neurogastroenterol Motil. 2014 May;26(5):705-14. doi: 10.1111/nmo.12320. Epub 2014 Mar 4. PMID 24588932